CLINICAL TRIAL: NCT03528694
Title: A Phase III Randomized, Open-Label, Multi-Center, Global Study of Durvalumab and Bacillus Calmette-Guerin (BCG) Administered as Combination Therapy Versus BCG Alone in High-Risk, BCG Naïve Non-Muscle Invasive Bladder Cancer Patients
Brief Title: Assessment of Efficacy and Safety of Durvalumab Plus BCG Compared to the Standard Therapy With BCG in Non-muscle Invasive Bladder Cancer
Acronym: POTOMAC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D419JC00001; 2017-002979-26 (EudraCT Number)
Record Dates: First submitted 2018-02-28; First posted 2018-05-18 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Non-muscle-invasive Bladder Cancer
Keywords: Durvalumab; BCG; MEDI4736; NMIBC; PD-L1; DFS; OS
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — durvalumab; BCG Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Durvalumab plus BCG (induction + maintenance) (Experimental): Durvalumab (MEDI4736) plus Bacillus Calmette-Guerrin (BCG) combination therapy
  Interventions: Biological: Durvalumab (MEDI4736); Biological: Bacillus Calmette-Guerin (BCG)
- Durvalumab plus BCG (induction only) (Experimental): Durvalumab (MEDI4736) plus Bacillus Calmette-Guerrin (BCG) combination therapy
  Interventions: Biological: Durvalumab (MEDI4736); Biological: Bacillus Calmette-Guerin (BCG)
- BCG treatment (Standard of care therapy) (Active Comparator): Bacillus Calmette-Guerrin (BCG) standard of care treatment
  Interventions: Biological: Bacillus Calmette-Guerin (BCG)

INTERVENTIONS:
Biological: Durvalumab (MEDI4736) — Investigational product
  Arms: Durvalumab plus BCG (induction + maintenance); Durvalumab plus BCG (induction only)
Biological: Bacillus Calmette-Guerin (BCG) — Standard of care

SUMMARY:
This is a randomized, open-label, multi-center, global, phase III study to determine the efficacy and safety of Durvalumab + BCG combination therapy in the treatment of patients with non-muscle-invasive bladder cancer

DETAILED DESCRIPTION:
Patients will be randomized in a 1:1:1 ratio to receive treatment with Durvalumab + BCG combination therapies, or Standard of Care (SoC) therapy.

ELIGIBILITY:
Inclusion Criteria: For inclusion in the study, patients should fulfill the following criteria:

* Aged at least 18 years
* BCG-naïve (patients who have not received prior intravesical BCG or who previously received but stopped BCG more than 3 years before study entry are eligible)
* Local histological confirmation (based on pathology report) of high-risk transitional cell carcinoma of the urothelium of the urinary bladder confined to the mucosa or submucosa. A high risk tumor is defined as one of the following

  * T1 tumor
  * High grade/ G3 tumor
  * CIS
  * Multiple and recurrent and large (with diameter of largest tumor ≥3 cm) tumors (all conditions must be met in this point)
* Complete resection of all Ta/T1 papillary disease prior to randomization, with the TURBT removing high-risk NMIBC performed not more than 4 months before randomization in the study. Patients with residual CIS after TURBT are eligible
* No prior radiotherapy for bladder cancer
* No prior exposure to immune-mediated therapy of cancer including, but not limited to, other anti CTLA-4, anti-PD-1, anti-PD-L1, and anti-programmed cell death ligand 2 antibodies. Patients who have been treated with anticancer vaccines will be excluded

Exclusion Criteria:

Patients should not enter the study if any of the following exclusion criteria are fulfilled:

* Evidence of muscle-invasive, locally advanced, metastatic, and/or extra vesical bladder cancer (ie, T2, T3, T4, and / or stage IV)
* Concurrent extravesical (ie, urethra, ureter, or renal pelvis), non-muscle-invasive transitional cell carcinoma of the urothelium
* Previous investigational product (IP) assignment in the present study
* Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for noncancer related conditions (eg, hormone replacement therapy) is acceptable. Chemotherapy for previous instances of NMIBC is acceptable.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the Study Physician
  * Patients with celiac disease controlled by diet alone
* History of another primary malignancy except for

  * Malignancy treated with curative intent and with no known active disease ≥ 2 years before the first dose of IP and of low potential risk for recurrence during the study period
  * Adequately treated nonmelanoma skin cancer or lentigo maligna withoutevidence of disease
  * Adequately treated CIS without evidence of disease
  * Prostate cancer (tumor/node/metastasis stage) of stage ≤ T2cN0M0 without biochemical recurrence or progression that in the opinion of the Investigator does not require active intervention
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (eg, computed tomography [CT] scan premedication)

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1018 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2028-10-03 (Estimated)

PRIMARY OUTCOMES:
The efficacy of Durvalumab + BCG (induction plus maintenance) combination therapy compared to SoC in terms of Disease free survival (DFS) in patients with NMIBC | Up to 4 years

SECONDARY OUTCOMES:
The efficacy of Durvalumab + BCG (induction plus maintenance) therapy compare to SoC in terms of DFS after 24 months of last subject's last dose of IP | Up to 4 years
Disease-related symptoms and HRQoL in patients with NMIBC treated with Durvalumab + BCG combination therapies compared to SoC and compared to each other using the EORTC QLQ-C30 questionnaire | Up to 4 years
  EORTC QLQ-C30 measures cancer patients' functioning (HRQoL) and symptoms for all cancer types and consists of functional, symptom and a global measure of health status scales
Patient-reported treatment tolerability using specific PRO CTCAE symptoms | Up to 4 years
The serum concentration of Durvalumab plus BCG combination therapies | Up to 4 years
The immunogenicity of Durvalumab when used in combination with BCG treatment assessed by descriptive summary of presence of ADAs | Up to 4 years
  Serum will be tested for the presence of anti-drug antibodies.
The efficacy of Durvalumab + BCG (induction plus maintenance) therapy compare to SoC in terms of OS | Up to 7 years
The efficacy of Durvalumab + BCG (induction plus maintenance) combination therapy compared to SoC in terms of time to muscle invasive bladder cancer and/or metastatic disease | Up to 7 years
The efficacy of Durvalumab + BCG (induction only) combination therapy compared to SoC in terms of DFS after 24 months of last subject's last dose of IP | Up to 4 years
The efficacy of Durvalumab + BCG combination therapies compared to each other in terms of DFS after 24 months of last subject's last dose of IP | Up to 4 years
The efficacy of Durvalumab + BCG (induction only) combination therapy compared to SoC in terms of OS | Up to 7 years
The efficacy of Durvalumab + BCG combination therapies compared to each other in terms of OS | Up to 7 years
The efficacy of Durvalumab + BCG (induction only) combination therapy compared to SoC in terms of time to muscle invasive bladder cancer and/or metastatic disease | Up to 7 years
The efficacy of Durvalumab + BCG combination therapies compared to each other in terms of time to muscle invasive bladder cancer and/or metastatic disease | Up to 7 years
Disease-related symptoms and HRQoL in patients with NMIBC treated with Durvalumab + BCG combination therapies compared to SoC and compared to each other using the the EORTC QLQ NMIBC24 questionnaire | Up to 4 years
  EORTC QLQ-NMIBC24 assesses disease-specific symptoms of patients with intermediate to high-risk NMIBC.
The efficacy of durvalumab + BCG combination therapy compared to SoC in terms of CRR for patients with CIS prior to study entry or at baseline cystoscopy | Up to 4 years
  CRR at 6 months in patients with CIS prior to the study entry or at baseline cystoscopy

OTHER OUTCOMES:
Number of treatment-related adverse events as assessed by CTCAE v4.0 in patients receiving Durvalumab + BCG combination therapies compared to SoC | Up to 4 years
  The safety and tolerability profile of Durvalumab + BCG combination therapies compared to SoC using vital signs, laboratory data, electrocardiograms (ECGs), and adverse event data.

CONTACTS AND LOCATIONS:
Locations (100):
- Australia (8):
  - Research Site, Auchenflower
  - Research Site, Box Hill
  - Research Site, Brisbane
  - Research Site, Kogarah
  - Research Site, Orange
  - Research Site, Parkville
  - Research Site, Westmead
  - Research Site, Wollongong
- Austria (5):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Linz
  - Research Site, Salzburg
  - Research Site, Vienna
- Belgium (4):
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Roeselare
- Canada (5):
  - Research Site, Kingston, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- France (8):
  - Research Site, Amiens
  - Research Site, Angers
  - Research Site, Bordeaux
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Strasbourg
  - Research Site, Suresnes
- Germany (14):
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Duisburg
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Marburg
  - Research Site, Mettmann
  - Research Site, Mühlheim An Der Ruhr
  - Research Site, München
  - Research Site, Münster
  - Research Site, Nürtingen
  - Research Site, Wesel
  - Research Site, Würselen
  - Research Site, Zirndorf
- Japan (19):
  - Research Site, Bunkyō City
  - Research Site, Fukuoka
  - Research Site, Hirosaki-shi
  - Research Site, Kanazawa
  - Research Site, Kita-gun
  - Research Site, Koshigaya-shi
  - Research Site, Kōtoku
  - Research Site, Matsuyama
  - Research Site, Miyazaki
  - Research Site, Nagasaki
  - Research Site, Nagoya
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Osakasayama-shi
  - Research Site, Sapporo
  - Research Site, Shinjuku-ku
  - Research Site, Toyama
  - Research Site, Tsukuba
  - Research Site, Yokohama
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Breda
  - Research Site, Utrecht
- Poland (8):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Grudziądz
  - Research Site, Koszalin
  - Research Site, Piotrkow Trybunalski
  - Research Site, Poznan
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Russia (9):
  - Research Site, Ivanovo
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Obninsk
  - Research Site, Omsk
  - Research Site, Saint Petersburg
  - Research Site, Vologda
  - Research Site, Yaroslavl
- Spain (10):
  - Research Site, Badajoz
  - Research Site, Barcelona
  - Research Site, Elche(Alicante)
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Oviedo
  - Research Site, Pamplona
  - Research Site, Pozuelo de Alarcón
  - Research Site, Seville
  - Research Site, Valencia
- United Kingdom (7):
  - Research Site, Birmingham
  - Research Site, Glasgow
  - Research Site, Guildford
  - Research Site, London
  - Research Site, Sheffield
  - Research Site, Southampton
  - Research Site, Taunton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] De Santis M, Palou Redorta J, Nishiyama H, Krawczynski M, Seyitkuliev A, Novikov A, Guerrero-Ramos F, Zukov R, Kato M, Kawahara T, Goeman L, Puente J, Hellmis E, Powles T, Radziszewski P, Gust KM, Vasey P, Bigot P, Fradet Y, Hunting J, Armstrong J, Boulos S, Hois S, Shore ND; POTOMAC Investigators. Durvalumab in combination with BCG for BCG-naive, high-risk, non-muscle-invasive bladder cancer (POTOMAC): final analysis of a randomised, open-label, phase 3 trial. Lancet. 2025 Nov 8;406(10516):2221-2234. doi: 10.1016/S0140-6736(25)01897-5. Epub 2025 Oct 17. PMID 41115436